CLINICAL TRIAL: NCT01689155
Title: Post-licensure Safety Surveillance Study of Menactra® Vaccine When Administered As a 2-dose Schedule to Children 9 Months Through 23 Months of Age.
Brief Title: Post-licensure Safety Surveillance Study of Menactra Vaccine When Administered As a 2-dose Schedule to Children
Status: Completed | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: MTA57; U 1111-1120-1574 (Other: WHO)
Record Dates: First submitted 2012-09-14; First posted 2012-09-21 (Estimated); Results first posted 2016-11-11 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-09

CONDITIONS: Meningitis; Meningococcal Infection
Keywords: Meningitis; Meningococcal Infection; Menactra®
MeSH Terms: conditions — Meningitis; Meningococcal Infections | interventions — Meningococcal Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Group: Participants must have received Menactra Vaccine according to routine clinical practice.
  Interventions: Biological: Menactra®: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate

INTERVENTIONS:
Biological: Menactra®: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate — 0.5 mL, Intramuscular
  Other Names: Menactra®

SUMMARY:
This is a passive-surveillance study that will accrue subjects for surveillance. For each accrued subject, surveillance for outcomes will continue for six months following the first dose. If a second dose is given within that time, then surveillance will be continued for six months following the second dose.

Observational Objective:

* To describe and characterize adverse events occurring after vaccination with Menactra vaccine.

DETAILED DESCRIPTION:
The study will be carried out in collaboration with the Kaiser Permanente Medical Care Program (KPMCP) under the direction of the Kaiser Permanente Vaccine Study Center (KPVSC). KPMCP is a closed-panel healthcare organization that maintains comprehensive encounter databases that capture all medical care received by enrollees.

Vaccination will be according to routine clinical practice. Vaccination databases will be reviewed to identify eligible persons receiving Menactra vaccine within the KPMCP system.

ELIGIBILITY:
Inclusion Criteria:

* Age 9 to 23 months at the time of receipt of the first dose of Menactra vaccine during the study period.

Ages: 9 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants at age 9 to 23 months at the time of receipt of the first dose of Menactra vaccine according to routine clinical practice during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2011-06; Primary Completion 2015-06 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (1):
- Oakland, California, United States

REFERENCES:
- [Derived] Hansen J, Zhang L, Eaton A, Baxter R, Robertson CA, Decker MD, Greenberg DP, Bassily E, Klein NP. Post-licensure safety surveillance study of routine use of quadrivalent meningococcal diphtheria toxoid conjugate vaccine (MenACWY-D) in infants and children. Vaccine. 2018 Apr 12;36(16):2133-2138. doi: 10.1016/j.vaccine.2018.02.107. Epub 2018 Mar 14. PMID 29550195
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participant accrual occurred from 16 June 2011 through 20 June 2014.
Pre-assignment Details: Databases of Kaiser Permanente in Northern California (KPNC) were reviewed to describe and characterize adverse events occurring after use of Menactra vaccine in routine clinical practice. Rates of events occurring in a risk window for participants were compared with rates of events occurring in a control window for the same participants.
Groups:
- Menactra Vaccine Recipients: Participants 9 months through 23 months of age receiving Menactra vaccine within the study institution following licensure of the vaccine for this age indication. KPNC databases were used; Menactra vaccine was administered according to routine clinical practice.
Period: Overall Study
Arm/Group | Menactra Vaccine Recipients
Started | 116
Completed | 116
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants age 9 months through 23 months of age receiving Menactra vaccine within the study institution following licensure of the vaccine for this age indication. KPNC databases were used; Menactra vaccine was administered according to routine clinical practice.
Arm/Group | Menactra Vaccine Recipients
Number analyzed (Participants) | 116
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 116
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 15.9 (5.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 55
Region of Enrollment [Number; unit: Participants]
  United States | 116
Seasonality [Number; unit: Participants] — Data represent participants receiving vaccine during time period shown. Four participants received 2 doses of Menactra; each dose is accounted for in the appropriate time period.
  Participants
    December - February | 30
    March - May | 39
    June - August | 22
    September - November | 29

OUTCOME MEASURES:

1. Primary Outcome: Rates of Safety Outcomes at Days 0-30 vs Days 31-75 After Menactra Vaccine - Emergency Room Database.
Description: Incidence rates for each event were calculated as the number of events divided by person-time and expressed as events per 1,000 person-months in each comparison widow. The risk window was Days 0-30 following vaccination; the control window was Days 31-75 post-vaccination.
Time Frame: Day 0 up to Day 75 post-vaccination
Population: Eligible participants who received Menactra vaccine during the study period and captured in the KPNC databases were included in the analysis.
Measure: Number; unit: Events per 1,000 person-months
Groups:
- Control Group: There was no separate control group per se. For all analyses, rates of events in a risk window for participants were compared with rates of events in a control window for the same participants.
Arm/Group | Menactra Vaccine Recipients | Control Group
Number analyzed (Participants) | 116 | 116
Events per 1,000 person-months
  Asthma | 0.009 | 0.006
  Cough | 0.009 | 0.006
  Febrile Seizure | 0.009 | 0.000
  Otitis Media | 0.009 | 0.000
  Trauma | 0.019 | 0.000
  Upper Respiratory Infection | 0.009 | 0.000
  Viral Syndrome | 0.009 | 0.000
  Vomiting (ER) | 0.009 | 0.000

2. Other Pre Specified Outcome: Rates of Safety Outcomes at Days 0-30 vs Days 31-75 After Menactra Vaccine - Hospital Database.
Description: Incidence rates for identified events were to be calculated as the number of events divided by person-time and expressed as events per 1,000 person-months in each comparison widow. The risk window was Days 0-30 following vaccination; the control window was Days 31-75 post-vaccination. Note: No events were identified in the hospital database.
Time Frame: Day 0 up to Day 75 post-vaccination
Population: All participants who received Menactra vaccine during the study period and captured in the KPNC databases were included in the analysis.
Measure: Number; unit: Events per 1,000 person-months
Arm/Group | Menactra Vaccine Recipients | Control Group
Number analyzed (Participants) | 116 | 116
Events per 1,000 person-months | 0 | 0

3. Other Pre Specified Outcome: Rates of Safety Outcomes at Days 0-30 vs Days 31-75 After Menactra Vaccine - Clinic Database.
Description: Incidence rates for pre-specified events were to be calculated as the number of events divided by person-time and expressed as events per 1,000 person-months in each comparison widow. The risk window was Days 0-30 following vaccination; the control window was Days 31-75 post-vaccination. Pre-specified neurological conditions, hypersensitivity reactions, and new-onset autoimmune disease were selected for monitoring in the clinical database. Note: None of these events were identified in the clinic database.
Time Frame: Day 0 up to Day 75 post-vaccination
Population: as for outcome 2
Measure: Number; unit: Events per 1,000 person-months
Arm/Group | Menactra Vaccine Recipients | Control Group
Number analyzed (Participants) | 116 | 116
Events per 1,000 person-months | 0 | 0

ADVERSE EVENTS:
Time Frame: Surveillance period for adverse events was from the day of vaccination to 6 months post-final vaccination, an average of 6 months.
Groups:
- Menactra Vaccine Recipients: Participants who received Menactra vaccine during the study period from the Kaiser Permanente databases.
Arm/Group | Menactra Vaccine Recipients
Serious Adverse Events (participants affected / at risk) | 0/116
Other Adverse Events (participants affected / at risk) | 0/116

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.